CLINICAL TRIAL: NCT02243306
Title: A Repeat-Dose, Open-Label, Parallel-Group Study to Assess the Pharmacokinetics of GSK1278863 and Metabolites in Subjects With End Stage Renal Disease Undergoing Peritoneal Dialysis
Brief Title: Study to Assess the Pharmacokinetics of GSK1278863 in Subjects With End Stage Renal Disease Undergoing Peritoneal Dialysis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 200942; 2014-001197-34 (EudraCT Number)
Record Dates: First submitted 2014-05-29; First posted 2014-09-17 (Estimated); Results first posted 2019-03-11 (Actual); Last update posted 2019-04-09 (Actual); Status verified 2019-03

CONDITIONS: Anaemia
Keywords: pharmacokinetics; Chronic kidney disease; peritoneal dialysis; hemoglobin; Anemia; GSK1278863; Prolyl hydroxylase inhibitor; erythropoiesis stimulating agents
MeSH Terms: conditions — Anemia; Renal Insufficiency, Chronic | interventions — GSK1278863

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1 (Experimental): Subjects on continuous ambulatory peritoneal dialysis (CAPD) will receive 5 mg of GSK1278863 orally, once daily for 14 days.
  Interventions: Drug: GSK1278863
- Cohort 2 (Experimental): Subjects on automated peritoneal dialysis (APD) will receive 5 mg of GSK1278863 orally, once daily for 14 days
  Interventions: Drug: GSK1278863

INTERVENTIONS:
Drug: GSK1278863 — Round, biconvex, white film coated tablet containing 5 mg GSK1278863.

SUMMARY:
GSK1278863 is an orally-active, novel small molecule agent which inhibits hypoxia-inducible factor (HIF) prolyl -4- hydroxylases (PHDs) and is in development for the treatment of anaemia associated with chronic kidney disease (CKD). As the kidney represents a major site of elimination for many drugs and their metabolites, and GSK1278863 will be administered to subjects with various stages of renal disease, it is important to characterize the pharmacokinetics in this target patient population. The purpose of this study is to characterize the pharmacokinetics of GSK1278863 and its metabolites in subjects with end stage renal disease (ESRD) undergoing peritoneal dialysis. This will be a repeat-dose, open-label, parallel-group study. Approximately 30 subjects with ESRD will be enrolled in two cohorts (15 subjects in each cohort) to ensure that 6 subjects on continuous ambulatory peritoneal dialysis (CAPD) (cohort 1) and 6 subjects on automated peritoneal dialysis APD (cohort 2) complete dosing and critical assessments. GSK1278863 will be administered once daily for 14 days. Primary pharmacokinetic assessments will be made on Days 1 and 14.

ELIGIBILITY:
Inclusion Criteria:

SAFETY:

* Satisfactory medical evaluation based upon medical history, medication history, physical examination, and clinical laboratory data obtained at the Screening visit. The determination of clinical significance will be made by the Investigator and the GlaxoSmithKline (GSK) Medical Monitor and will require that the finding is unlikely to introduce additional risk factors or interfere with the study procedures, or the integrity of the study.
* Corrected QT interval (QTc) <470 milliseconds (msec) OR QTc <480 msec in subjects with Bundle Branch Block. These should be based on average of triplicate values obtained over a brief recording period at Screening and on Day -1 and the single reading on Day 17. The same QT correction formula should be used to determine inclusion and discontinuation for any individual subject throughout the study.
* Vitamin B12 and folate above the lower limit of normal at Screening.
* Aspartate aminotransferase (AST), Alanine aminotransferase (ALT), and bilirubin <=1.5 x upper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).

EFFICACY:

* A subject is eligible to enroll and participate in this study if he/she has ESRD and is on peritoneal dialysis for at least 2 months with an average urine output of <750 mL/daily with a combined weekly (urine and peritoneal dialysis output) Kt/V urea >1.7 measured at any time within last 3 months.
* No history of peritoneal dialysis-associated peritonitis, peritoneal catheter tunnel (exit site) infection or leakage for at least 3 months before study.
* Meets the following erythropoiesis stimulating agent (ESA) criteria: Is ESA naive (i.e., no ESA use within the previous 12 weeks of screening) OR agrees to discontinue ESA (if currently using ESA) for at least 7 days prior to first dose of GSK1278863 until completion of Follow-up visit (If the subject has a scheduled ESA interval which is <=7 days, ESA treatment must be discontinued for at least 7 days prior to first dose of GSK1278863. If the subject has a scheduled ESA interval which is >7 days, ESA treatment must be discontinued for at least the scheduled interval length [e.g., if ESA interval is 14 days, then ESA must be discontinued for >=14 days] prior to the first dose of GSK1278863)
* Has a haemoglobin value: For ESA naïve subjects: <10.0 g/dL (UK site(s) only: <=11.0 g/dL); For subjects receiving ongoing ESA treatment: <=11.0 g/dL at Screening (UK site(s) only: <=12.0 g/dL at Screening).

OTHER:

* Subjects who are >=18 years of age at the time of Screening.
* A female subject is eligible to participate if she is of: (a) Childbearing potential, and agrees to use one of the contraception methods described in the protocol. This criterion must be followed from the time of Screening until completion of the Follow-up Visit; (b) Non-childbearing potential, defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea (In questionable cases, a blood sample with simultaneous follicle stimulating hormone (FSH) 23.0-116.3 international units (IU)/litre (L) and estradiol <=10 picograms (pg)/mL (or <=37 picomoles [pmol]/L) is confirmatory). Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods described in the protocol if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment. For most forms of HRT, at least 2 months must elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method.
* Body weight >45 kilograms (kg) and <140 kg at Screening.
* The subject is mentally and legally able to comply with the requirements and restrictions of the protocol and has provided signed informed consent prior to participation in any protocol-specific procedures, including Screening procedures.

Exclusion Criteria:

SAFETY

* A positive test for Human Immunodeficiency Virus (HIV) antibody.
* Uncontrolled hypertension (diastolic blood pressure [BP] >100 millimetres of mercury [mmHg] or systolic BP >170 mmHg) at Screening.
* History of drug abuse or dependence within 6 months of the study.
* History of sensitivity to GSK1278863, or its components thereof or a history of drug or other allergy that, in the opinion of the Investigator or GSK Medical Monitor, contraindicates their participation.
* History of sensitivity to heparin or heparin-induced thrombocytopenia (if the clinical research unit uses heparin to maintain intravenous cannula patency).
* History of thrombosis defined as deep vein thrombosis, stroke, pulmonary embolism or other thrombosis related condition within 3 months prior to Screening.
* History of myocardial infarction or acute coronary syndrome within 3 months prior to Screening.
* History of stroke or transient ischaemic attack within 3 months prior to Screening.
* Subjects with a pre-existing condition interfering with normal gastrointestinal anatomy or motility, and/or hepatic function that could interfere with the absorption, metabolism, and/or excretion of GSK1278863. Examples of conditions that could interfere with normal gastrointestinal anatomy or motility include gastrointestinal bypass surgery, partial or total gastrectomy, small bowel resection, vagotomy, malabsorption, Crohn's disease, ulcerative colitis, or celiac sprue. Examples of conditions that could interfere with hepatic function include Gilbert's syndrome.
* Evidence of active peptic, duodenal or esophageal ulcer disease at Screening OR history of clinically significant gastro-intestinal (GI) bleeding within 3 months prior to Screening.
* Subjects with chronic inflammatory disease that could impact erythropoiesis (e.g. scleroderma, systemic lupus erythematosis, rheumatoid arthritis, celiac disease).
* Subjects with a history of symptomatic right heart failure.
* Subjects with Class III or Class IV heart failure, as defined by the New York Heart Association (NYHA) functional classification system.
* Active malignancy or diagnosis of malignancy within 5 years prior to Screening (excluding successfully treated basal or squamous cell carcinoma).
* History of proliferative vascular eye disease (e.g., choroidal or retinal disease, such as neovascular age-related macular degeneration, proliferative diabetic retinopathy or macular edema) based upon having had an ophthalmologic exam within 12 months prior to the end of the Screening period (The screening period is from the screening visit until Day -1).
* Pregnant females as determined by positive serum human chorionic gonadotropin (hCG) test at Screening or Day -1.
* Lactating females.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period prior to first dose.
* Consumption of red wine, grapefruit (juice), blood orange (juice), star fruit, onions, kale, broccoli, green beans, or apples from 7 days prior to the first dose of investigational product until the Follow-up visit, unless in the opinion of the Investigator and GSK Medical Monitor this will not interfere with the study procedures and compromise subject safety.
* Use or planned use of any prescription or non-prescription drugs that are prohibited within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of GSK1278863 until completion of the follow-up visit, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* The following medications are specifically prohibited for the duration of the study (from Screening to the follow-up visit at the end of the study): Chronic use of non-steroidal anti-inflammatory drugs (NSAIDs) with the exception of low dose (<=325 mg/day) aspirin/acetylsalicylic acid. Occasional NSAID use is permitted; Immunosuppressant drugs and drugs used to treat malignancies (including corticosteroids at doses >10 mg prednisolone per day or equivalent) within 2 weeks of first dose of GSK1278863. Note: Failed transplant subjects back on peritoneal dialysis are eligible for participating in this study but should not be on immunosuppressive medications within 3 months prior to Screening.
* The subject has participated in a clinical trial and has received an experimental investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).

EFFICACY:

* The values of ferritin and transferrin within 3 months prior to Screening are: (a) transferrin saturation <20%; (b) serum ferritin <100 micrograms (mcg)/L

OTHER:

* A positive pre-dosing drug/alcohol screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines. A positive pre-dosing screen for medications that are prescribed to a renal subject for pre-existing condition(s), may be allowed if in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of >21 units for males or >14 units for females. One unit is equivalent to 8 g of alcohol: a half-pint (approximately240 mL) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits.
* History of regular use within 6 months of the study of tobacco- or nicotine-containing products in excess of 20 cigarettes per day or equivalent.
* Unwillingness or inability to follow the procedures, or lifestyle and/or dietary restrictions outlined in the informed consent and as directed by site staff.
* Subject is either an immediate family member of a participating Investigator, study coordinator, employee of an Investigator; or is a member of the staff conducting the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-10-24 (Actual); Primary Completion 2017-05-10 (Actual); Study Completion 2017-05-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- United States (2):
  - GSK Investigational Site, Lakewood, Colorado
  - GSK Investigational Site, Minneapolis, Minnesota

REFERENCES:
- [Background] Caltabiano S, Cizman B, Burns O, Mahar KM, Johnson BM, Ramanjineyulu B, Serbest G, Cobitz AR. Effect of renal function and dialysis modality on daprodustat and predominant metabolite exposure. Clin Kidney J. 2019 Feb 18;12(5):693-701. doi: 10.1093/ckj/sfz013. eCollection 2019 Oct. PMID 31583094

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This repeat-dose, pharmacokinetic (PK) study of GSK1278863 was conducted at two centers in the United States (US). Participants with End Stage Renal Disease (ESRD) undergoing continuous ambulatory peritoneal dialysis (CAPD) or automated peritoneal dialysis (APD) were included in this study.
Pre-assignment Details: A total of 20 participants with ESRD were screened; of which 12 were screen failures and 8 entered the study to receive 5 milligrams (mg) of GSK1278863 once daily for 14 days.
Groups:
- Participants Undergoing CAPD: Participants on CAPD received 1 tablet (5 mg) of GSK1278863 by oral route once daily with half glass of water for 14 days. On Day 1 and Day 14, the dose was administered within 30 minutes after completion of night CAPD treatment or morning last fill of peritoneal dialysis fluid; on any other study days, the dose was administered within 2 hours after completion of night CAPD treatment or morning last fill of peritoneal dialysis fluid.
- Participants Undergoing APD: Participants on APD received 1 tablet (5 mg) of GSK1278863 by oral route once daily with half glass of water for 14 days. On Day 1 and Day 14, the dose was administered within 30 minutes after completion of night APD treatment or morning last fill of peritoneal dialysis fluid; on any other study days, the dose was administered within 2 hours after completion of night APD treatment or morning last fill of peritoneal dialysis fluid.
Period: Overall Study
Arm/Group | Participants Undergoing CAPD | Participants Undergoing APD
Started | 1 | 7
Completed | 1 | 4
Not Completed | 0 | 3
Not completed — Adverse Event | 0 | 1
Not completed — Other: Reached stopping criteria | 0 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Participants Undergoing CAPD: Participants on CAPD received 1 tablet (5 mg) of GSK1278863 by oral route once daily with half glass of water for 14 days. On Day 1 and Day14, the dose was administered within 30 minutes after completion of night CAPD treatment or morning last fill of peritoneal dialysis fluid; on any other study days, the dose was administered within 2 hours after completion of night CAPD treatment or morning last fill of peritoneal dialysis fluid.
- Participants Undergoing APD: Participants on APD received 1 tablet (5 mg) of GSK1278863 by oral route once daily with half glass of water for 14 days. On Day 1 and Day14, the dose was administered within 30 minutes after completion of night APD treatment or morning last fill of peritoneal dialysis fluid; on any other study days, the dose was administered within 2 hours after completion of night APD treatment or morning last fill of peritoneal dialysis fluid.
- Total: Total of all reporting groups
Arm/Group | Participants Undergoing CAPD | Participants Undergoing APD | Total
Number analyzed (Participants) | 1 | 7 | 8
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age is calculated based on screening date, using date of birth, truncated to integer value.
  Years | 44.0 (NA) — Standard deviation could not be calculated for CAPD arm due to low number of participants | 57.4 (12.01) | 55.8 (12.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2
  Male | 1 | 5 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race customized: American Indian or Alaska Native Heritage | 0 | 1 | 1
  Race customized: Black or African American Heritage | 0 | 3 | 3
  Race customized: White- White/Caucasian/European Heritage | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve (AUC) Over the Dosing Interval (AUC[0-tau]) of GSK1278863 and Its Metabolites
Description: Serial blood samples were collected from participants at indicated time points for Pharmacokinetic (PK) analysis of GSK1278863 and its metabolites (GSK2391220, GSK2487818, GSK2506102, GSK2531398, GSK2531403 and GSK2531401). Geometric mean and geometric coefficient of variation has been presented for all metabolites. NA indicates data is not available. Geometric coefficient of variation could not be calculated for CAPD cohort due to small number of participants. PK Population comprised of participants in the 'All Subjects' Population for whom a PK sample was obtained and analyzed.
Time Frame: Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24 hours post-dose on Day 1; Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 48, 72 hours post-dose on Day 14
Population: PK Population. Only those participants available at the specified time points were analyzed (represented by n=x in category titles).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour into nanograms per milliliter
Arm/Group | Participants Undergoing CAPD | Participants Undergoing APD
Number analyzed (Participants) | 1 | 7
Hour into nanograms per milliliter
  GSK1278863; Day 1; n=1, 7 | 184.9863 (NA) — Geometric coefficient of variation could not be calculated for CAPD cohort due to small number of participants. | 138.6511 (93.5)
  GSK1278863; Day 14; n=1, 4: number analyzed (Participants) | 1 | 4
  GSK1278863; Day 14; n=1, 4 | 162.9366 (NA) — Geometric coefficient of variation could not be calculated for CAPD cohort due to small number of participants. | 131.2826 (78.8)
  GSK2391220; Day 1; n=1, 7 | 245.8999 (NA) — Geometric coefficient of variation could not be calculated for CAPD cohort due to small number of participants. | 147.8039 (47.7)
  GSK2391220; Day 14; n=1, 4: number analyzed (Participants) | 1 | 4
  GSK2391220; Day 14; n=1, 4 | 258.1199 (NA) — Geometric coefficient of variation could not be calculated for CAPD cohort due to small number of participants. | 162.0324 (50.7)
  GSK2487818; Day 1; n=1, 7 | 116.2608 (NA) — Geometric coefficient of variation could not be calculated for CAPD cohort due to small number of participants. | 67.4130 (39.1)
  GSK2487818; Day 14; n=1, 4: number analyzed (Participants) | 1 | 4
  GSK2487818; Day 14; n=1, 4 | 114.1857 (NA) — Geometric coefficient of variation could not be calculated for CAPD cohort due to small number of participants. | 59.6501 (51.5)
  GSK2506102; Day 1; n=1,6: number analyzed (Participants) | 1 | 6
  GSK2506102; Day 1; n=1,6 | 59.0619 (NA) — Geometric coefficient of variation could not be calculated for CAPD cohort due to small number of participants. | 44.8180 (37.8)
  GSK2506102; Day 14; n=1, 4: number analyzed (Participants) | 1 | 4
  GSK2506102; Day 14; n=1, 4 | 82.9794 (NA) — Geometric coefficient of variation could not be calculated for CAPD cohort due to small number of participants. | 65.2188 (63.0)
  GSK2531398; Day 1; n=1, 7 | 97.0339 (NA) — Geometric coefficient of variation could not be calculated for CAPD cohort due to small number of participants. | 63.0979 (45.5)
  GSK2531398; Day 14; n=1, 4: number analyzed (Participants) | 1 | 4
  GSK2531398; Day 14; n=1, 4 | 97.6587 (NA) — Geometric coefficient of variation could not be calculated for CAPD cohort due to small number of participants. | 65.9664 (53.5)
  GSK2531403; Day 1; n=1, 7 | 291.3067 (NA) — Geometric coefficient of variation could not be calculated for CAPD cohort due to small number of participants. | 170.4958 (45.5)
  GSK2531403; Day 14; n=1, 4: number analyzed (Participants) | 1 | 4
  GSK2531403; Day 14; n=1, 4 | 360.2268 (NA) — Geometric coefficient of variation could not be calculated for CAPD cohort due to small number of participants. | 228.6081 (69.4)
  GSK2531401; Day 1; n=1, 6: number analyzed (Participants) | 1 | 6
  GSK2531401; Day 1; n=1, 6 | 173.5919 (NA) — Geometric coefficient of variation could not be calculated for CAPD cohort due to small number of participants. | 104.2971 (48.6)
  GSK2531401; Day 14; n=1, 4: number analyzed (Participants) | 1 | 4
  GSK2531401; Day 14; n=1, 4 | 242.0514 (NA) — Geometric coefficient of variation could not be calculated for CAPD cohort due to small number of participants. | 205.7281 (20.1)

2. Primary Outcome: AUC From Time Zero (Pre-dose) Extrapolated to Infinite Time (AUC [0-inf]) of GSK1278863 and Its Metabolites
Description: Serial blood samples were collected from participants at indicated time points for PK analysis of GSK1278863 and its metabolites (GSK2487818 and GSK2531398). Geometric mean and geometric coefficient of variation has been presented for all metabolites. NA indicates data is not available. Geometric coefficient of variation could not be calculated for CAPD cohort due to small number of participants.
Time Frame: Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24 hours post-dose on Day 1
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour into nanograms per milliliter
Arm/Group | Participants Undergoing CAPD | Participants Undergoing APD
Number analyzed (Participants) | 1 | 7
Hour into nanograms per milliliter
  GSK1278863 | 184.9888 (NA) — Geometric coefficient of variation could not be calculated for CAPD cohort due to small number of participants. | 138.6860 (93.6)
  GSK2487818 | 117.2111 (NA) — Geometric coefficient of variation could not be calculated for CAPD cohort due to small number of participants. | 68.5089 (39.9)
  GSK2531398 | 104.5268 (NA) — Geometric coefficient of variation could not be calculated for CAPD cohort due to small number of participants. | 73.9865 (51.3)

3. Primary Outcome: Maximum Observed Concentration (Cmax) of GSK1278863 and Its Metabolites
Description: Serial blood samples were collected from participants at indicated time points for PK analysis of GSK1278863 and its metabolites (GSK2391220, GSK2487818, GSK2506102, GSK2531398, GSK2531403 and GSK2531401). Geometric mean and geometric coefficient of variation has been presented for all metabolites. NA indicates data is not available. Geometric coefficient of variation could not be calculated for CAPD cohort due to small number of participants. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Participants Undergoing CAPD | Participants Undergoing APD
Number analyzed (Participants) | 1 | 7
Nanograms per milliliter
  GSK1278863; Day 1; n= 1, 7 | 90.400 (NA) — Geometric coefficient of variation could not be calculated for CAPD cohort due to small number of participants. | 58.771 (96.7)
  GSK1278863; Day 14; n= 1, 4: number analyzed (Participants) | 1 | 4
  GSK1278863; Day 14; n= 1, 4 | 57.800 (NA) — Geometric coefficient of variation could not be calculated for CAPD cohort due to small number of participants. | 30.303 (104.4)
  GSK2391220; Day 1; n= 1, 7 | 19.900 (NA) — Geometric coefficient of variation could not be calculated for CAPD cohort due to small number of participants. | 11.360 (44.3)
  GSK2391220; Day 14; n= 1, 4: number analyzed (Participants) | 1 | 4
  GSK2391220; Day 14; n= 1, 4 | 20.500 (NA) — Geometric coefficient of variation could not be calculated for CAPD cohort due to small number of participants. | 10.966 (33.1)
  GSK2487818; Day 1; n= 1, 7 | 19.400 (NA) — Geometric coefficient of variation could not be calculated for CAPD cohort due to small number of participants. | 10.117 (25.7)
  GSK2487818; Day 14; n= 1, 4: number analyzed (Participants) | 1 | 4
  GSK2487818; Day 14; n= 1, 4 | 18.400 (NA) — Geometric coefficient of variation could not be calculated for CAPD cohort due to small number of participants. | 7.262 (40.4)
  GSK2506102; Day 1; n= 1, 7 | 3.820 (NA) — Geometric coefficient of variation could not be calculated for CAPD cohort due to small number of participants. | 2.553 (42.7)
  GSK2506102; Day 14; n= 1, 4: number analyzed (Participants) | 1 | 4
  GSK2506102; Day 14; n= 1, 4 | 5.050 (NA) — Geometric coefficient of variation could not be calculated for CAPD cohort due to small number of participants. | 3.590 (46.5)
  GSK2531398; Day 1; n= 1, 7 | 9.300 (NA) — Geometric coefficient of variation could not be calculated for CAPD cohort due to small number of participants. | 5.370 (44.2)
  GSK2531398; Day 14; n= 1, 4: number analyzed (Participants) | 1 | 4
  GSK2531398; Day 14; n= 1, 4 | 9.220 (NA) — Geometric coefficient of variation could not be calculated for CAPD cohort due to small number of participants. | 4.857 (35.6)
  GSK2531403; Day 1; n= 1, 7 | 18.600 (NA) — Geometric coefficient of variation could not be calculated for CAPD cohort due to small number of participants. | 11.186 (36.7)
  GSK2531403; Day 14; n= 1, 4: number analyzed (Participants) | 1 | 4
  GSK2531403; Day 14; n= 1, 4 | 23.400 (NA) — Geometric coefficient of variation could not be calculated for CAPD cohort due to small number of participants. | 13.267 (48.2)
  GSK2531401; Day 1; n= 1, 7 | 9.920 (NA) — Geometric coefficient of variation could not be calculated for CAPD cohort due to small number of participants. | 4.715 (78.4)
  GSK2531401; Day 14; n= 1, 4: number analyzed (Participants) | 1 | 4
  GSK2531401; Day 14; n= 1, 4 | 13.300 (NA) — Geometric coefficient of variation could not be calculated for CAPD cohort due to small number of participants. | 10.404 (17.4)

4. Secondary Outcome: Number of Participants With Non-serious Adverse Events (AEs) and Serious AEs (SAEs)
Description: An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability, is a congenital anomaly/birth defect, other situations, and is associated with liver injury and impaired liver function. Analysis was performed on All Subjects Population which comprised of all enrolled participants who received at least one dose of study treatment.
Time Frame: Up to Day 24
Population: All subjects Population
Measure: Number; unit: Participants
Arm/Group | Participants Undergoing CAPD | Participants Undergoing APD
Number analyzed (Participants) | 1 | 7
Participants
  Non-serious AEs | 1 | 5
  SAEs | 0 | 0

5. Secondary Outcome: Change From Baseline in Glucose, Calcium, Chloride, Carbon-dioxide (CO2), Potassium, Sodium and Urea Levels
Description: Blood samples were collected from participants to evaluate clinical chemistry parameters including glucose, calcium, chloride, CO2, potassium, sodium and urea. Change from Baseline in clinical chemistry parameters at Day 17 are presented. Day-1 was considered as Baseline value. Change from Baseline was calculated as post-randomization values minus Baseline value. Mean and standard deviation are presented. NA indicates data is not available. Standard deviation could not be calculated for CAPD cohort due to small number of participants. Only participants with data available at the specified time point were analyzed.
Time Frame: Baseline and Day 17
Population: All Subjects Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Participants Undergoing CAPD | Participants Undergoing APD
Number analyzed (Participants) | 1 | 4
Millimoles per liter
  Glucose | -0.10 (NA) — Standard deviation could not be calculated for CAPD cohort due to small number of participants. | 0.27 (7.191)
  Calcium | 0.360 (NA) — Standard deviation could not be calculated for CAPD cohort due to small number of participants. | 0.040 (0.2026)
  Chloride | -2.0 (NA) — Standard deviation could not be calculated for CAPD cohort due to small number of participants. | -1.3 (2.99)
  CO2 | 0.0 (NA) — Standard deviation could not be calculated for CAPD cohort due to small number of participants. | 0.3 (5.19)
  Potassium | 0.20 (NA) — Standard deviation could not be calculated for CAPD cohort due to small number of participants. | -0.45 (0.580)
  Sodium | 2.0 (NA) — Standard deviation could not be calculated for CAPD cohort due to small number of participants. | -1.5 (3.70)
  Urea | 12.50 (NA) — Standard deviation could not be calculated for CAPD cohort due to small number of participants. | -0.38 (3.568)

6. Secondary Outcome: Change From Baseline in Albumin and Protein Levels
Description: Blood samples were collected from participants to evaluate clinical chemistry parameters including albumin and protein. Change from Baseline in clinical chemistry parameters at Day 17 are presented. Day-1 was considered as Baseline value. Change from Baseline was calculated as post-randomization values minus Baseline value. Mean and standard deviation are presented. NA indicates data is not available. Standard deviation could not be calculated for CAPD cohort due to small number of participants. Only participants with data available at the specified time point were analyzed.
Time Frame: Baseline and Day 17
Population: All Subjects Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Gram per liter (g/L)
Arm/Group | Participants Undergoing CAPD | Participants Undergoing APD
Number analyzed (Participants) | 1 | 4
Gram per liter (g/L)
  Albumin | 3.0 (NA) — Standard deviation could not be calculated for CAPD cohort due to small number of participants. | -1.3 (3.20)
  Protein | 5.0 (NA) — Standard deviation could not be calculated for CAPD cohort due to small number of participants. | -2.0 (5.48)

7. Secondary Outcome: Change From Baseline in Direct Bilirubin, Bilirubin, Creatinine and Urate Levels
Description: Blood samples were collected from participants to evaluate clinical chemistry parameters including direct bilirubin, bilirubin, creatinine and urate. Change from Baseline in clinical chemistry parameters at Day 17 are presented. Day-1 was considered as Baseline value. Change from Baseline was calculated as post-randomization values minus Baseline value. Mean and standard deviation are presented. NA indicates data is not available. Standard deviation could not be calculated for CAPD cohort due to small number of participants. Only participants with data available at the specified time point were analyzed.
Time Frame: Baseline and Day 17
Population: All Subjects Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Participants Undergoing CAPD | Participants Undergoing APD
Number analyzed (Participants) | 1 | 4
Micromoles per liter
  Direct bilirubin | 0.0 (NA) — Standard deviation could not be calculated for CAPD cohort due to small number of participants. | -0.5 (1.91)
  Bilirubin | -2.0 (NA) — Standard deviation could not be calculated for CAPD cohort due to small number of participants. | 0.5 (1.00)
  Creatinine | 13.30 (NA) — Standard deviation could not be calculated for CAPD cohort due to small number of participants. | -119.12 (312.679)
  Urate | -30.0 (NA) — Standard deviation could not be calculated for CAPD cohort due to small number of participants. | -25.0 (87.37)

8. Secondary Outcome: Change From Baseline in Alkaline Phosphatase (ALP), Aspartate Aminotransferase (AST) and Gamma Glutamyl Aminotransferase (GGT) Levels
Description: Blood samples were collected from participants to evaluate clinical chemistry parameters including ALP, AST and GGT. Change from Baseline in clinical chemistry parameters at Day 17 are presented. Day-1 was considered as Baseline value. Change from Baseline was calculated as post-randomization values minus Baseline value. Mean and standard deviation are presented. NA indicates data is not available. Standard deviation could not be calculated for CAPD cohort due to small number of participants. Only participants with data available at the specified time point were analyzed.
Time Frame: Baseline and Day 17
Population: All Subjects Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: International unit per liter (IU/L)
Arm/Group | Participants Undergoing CAPD | Participants Undergoing APD
Number analyzed (Participants) | 1 | 4
International unit per liter (IU/L)
  ALP | 5.0 (NA) — Standard deviation could not be calculated for CAPD cohort due to small number of participants. | -0.5 (16.52)
  AST | -1.0 (NA) — Standard deviation could not be calculated for CAPD cohort due to small number of participants. | -3.3 (3.77)
  GGT | 0.0 (NA) — Standard deviation could not be calculated for CAPD cohort due to small number of participants. | -6.3 (8.77)

9. Secondary Outcome: Change From Baseline in Alanine Aminotransferase (ALT) and Creatinine Kinase Levels
Description: Blood samples were collected from participants to evaluate clinical chemistry parameters including ALT and creatinine kinase. Change from Baseline in clinical chemistry parameters at Day 3, Day 7, Day 11, Day 14 and Day 17 are presented. Day-1 was considered as Baseline value. Change from Baseline was calculated as post-randomization values minus Baseline value. Mean and standard deviation are presented. NA indicates data is not available. Standard deviation could not be calculated for CAPD cohort due to small number of participants. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Baseline and Day 3, 7, 11, 14, 17
Population: All Subjects Population. Only those participants available at the specified time points were analyzed (represented by n=x in category titles).
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Participants Undergoing CAPD | Participants Undergoing APD
Number analyzed (Participants) | 1 | 7
IU/L
  ALT; Day 3; n= 1, 6: number analyzed (Participants) | 1 | 6
  ALT; Day 3; n= 1, 6 | -3.0 (NA) — Standard deviation could not be calculated for CAPD cohort due to small number of participants. | -0.7 (3.98)
  ALT; Day 7; n= 1, 4: number analyzed (Participants) | 1 | 4
  ALT; Day 7; n= 1, 4 | -7.0 (NA) — Standard deviation could not be calculated for CAPD cohort due to small number of participants. | -2.5 (5.32)
  ALT; Day 11; 1, 4: number analyzed (Participants) | 1 | 4
  ALT; Day 11; 1, 4 | -9.0 (NA) — Standard deviation could not be calculated for CAPD cohort due to small number of participants. | -3.5 (5.80)
  ALT; Day 14; n= 1, 4: number analyzed (Participants) | 1 | 4
  ALT; Day 14; n= 1, 4 | -7.0 (NA) — Standard deviation could not be calculated for CAPD cohort due to small number of participants. | -0.8 (3.86)
  ALT; Day 17; n= 1, 4: number analyzed (Participants) | 1 | 4
  ALT; Day 17; n= 1, 4 | -7.0 (NA) — Standard deviation could not be calculated for CAPD cohort due to small number of participants. | -1.0 (6.06)
  Creatine kinase; Day 3; n= 1, 6: number analyzed (Participants) | 1 | 6
  Creatine kinase; Day 3; n= 1, 6 | -12.0 (NA) — Standard deviation could not be calculated for CAPD cohort due to small number of participants. | -99.7 (161.17)
  Creatine kinase; Day 7; n= 1, 4: number analyzed (Participants) | 1 | 4
  Creatine kinase; Day 7; n= 1, 4 | -12.0 (NA) — Standard deviation could not be calculated for CAPD cohort due to small number of participants. | -137.8 (230.33)
  Creatine kinase; Day 11; n= 1, 4: number analyzed (Participants) | 1 | 4
  Creatine kinase; Day 11; n= 1, 4 | 1.0 (NA) — Standard deviation could not be calculated for CAPD cohort due to small number of participants. | -135.8 (273.85)
  Creatine kinase; Day 14; n= 1, 4: number analyzed (Participants) | 1 | 4
  Creatine kinase; Day 14; n= 1, 4 | 9.0 (NA) — Standard deviation could not be calculated for CAPD cohort due to small number of participants. | -183.5 (247.13)
  Creatine kinase; Day 17; n= 1, 4: number analyzed (Participants) | 1 | 4
  Creatine kinase; Day 17; n= 1, 4 | -2.0 (NA) — Standard deviation could not be calculated for CAPD cohort due to small number of participants. | -201.5 (191.83)

10. Secondary Outcome: Change From Baseline in Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils, Platelets and Leukocytes Levels
Description: Blood samples were collected from participants to evaluate clinical hematology parameters including basophils, eosinophils, lymphocytes, monocytes, neutrophils, platelets and leukocytes. Change from Baseline in clinical hematology parameters at Day 17 are presented. Day-1 was considered as Baseline value. Change from Baseline was calculated as post-randomization values minus Baseline value. NA indicates data is not available. Mean and standard deviation are presented. Standard deviation could not be calculated for CAPD cohort due to small number of participants. Only participants with data available at the specified time point were analyzed.
Time Frame: Baseline and Day 17
Population: All Subjects Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: 10^9 cells/liter
Arm/Group | Participants Undergoing CAPD | Participants Undergoing APD
Number analyzed (Participants) | 1 | 4
10^9 cells/liter
  Basophils | -0.020 (NA) — Standard deviation could not be calculated for CAPD cohort due to small number of participants. | 0.010 (0.0200)
  Eosinophils | -0.010 (NA) — Standard deviation could not be calculated for CAPD cohort due to small number of participants. | 0.060 (0.0804)
  Lymphocytes | 0.260 (NA) — Standard deviation could not be calculated for CAPD cohort due to small number of participants. | -0.138 (0.3974)
  Monocytes | 0.230 (NA) — Standard deviation could not be calculated for CAPD cohort due to small number of participants. | 0.060 (0.3389)
  Neutrophils | 1.350 (NA) — Standard deviation could not be calculated for CAPD cohort due to small number of participants. | -0.365 (1.1957)
  Platelets | 42.0 (NA) — Standard deviation could not be calculated for CAPD cohort due to small number of participants. | -21.0 (35.92)
  Leukocytes | 1.80 (NA) — Standard deviation could not be calculated for CAPD cohort due to small number of participants. | -0.35 (1.008)

11. Secondary Outcome: Change From Baseline in Erythrocyte and Reticulocyte Levels
Description: Blood samples were collected from participants to evaluate clinical hematology parameters including erythrocyte and reticulocyte. Change from Baseline in clinical hematology parameters at Day 17 are presented. Day-1 was considered as Baseline value. Change from Baseline was calculated as post-randomization values minus Baseline value. NA indicates data is not available. Mean and standard deviation are presented. Standard deviation could not be calculated for CAPD cohort due to small number of participants. Only participants with data available at the specified time point were analyzed.
Time Frame: Baseline and Day 17
Population: All Subjects Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: 10^12 cells/liter
Arm/Group | Participants Undergoing CAPD | Participants Undergoing APD
Number analyzed (Participants) | 1 | 4
10^12 cells/liter
  Erythrocytes | 0.00 (NA) — Standard deviation could not be calculated for CAPD cohort due to small number of participants. | -0.05 (0.412)
  Reticulocytes | 0.02840 (NA) — Standard deviation could not be calculated for CAPD cohort due to small number of participants. | -0.00165 (0.044431)

12. Secondary Outcome: Change From Baseline in Hematocrit Levels
Description: Blood samples were collected from participants to evaluate clinical hematology parameters including hematocrit. Change from Baseline in clinical hematology parameters at Day 17 are presented. Day-1 was considered as Baseline value. Change from Baseline was calculated as post-randomization values minus Baseline value. Mean and standard deviation are presented. NA indicates data is not available. Standard deviation could not be calculated for CAPD cohort due to small number of participants. Only participants with data available at the specified time point were analyzed.
Time Frame: Baseline and Day 17
Population: All Subjects Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | Participants Undergoing CAPD | Participants Undergoing APD
Number analyzed (Participants) | 1 | 4
Proportion of red blood cells in blood | 0.0070 (NA) — Standard deviation could not be calculated for CAPD cohort due to small number of participants. | -0.0100 (0.03880)

13. Secondary Outcome: Change From Baseline in Hemoglobin Levels
Description: Blood samples were collected from participants to evaluate clinical hematology parameters including hemoglobin. Change from Baseline in clinical hematology parameters at Day 3, Day 7, Day 11 and Day 17 are presented. Day-1 was considered as Baseline value. Change from Baseline was calculated as post-randomization values minus Baseline value. Mean and standard deviation are presented. NA indicates data is not available. Standard deviation could not be calculated for CAPD cohort due to small number of participants. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Baseline and Day 3, 7, 11, 17
Population: All Subjects Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Participants Undergoing CAPD | Participants Undergoing APD
Number analyzed (Participants) | 1 | 7
g/L
  Day 3; n= 1, 7 | 7.0 (NA) — Standard deviation could not be calculated for CAPD cohort due to small number of participants. | 3.1 (11.96)
  Day 7; n= 1, 5: number analyzed (Participants) | 1 | 5
  Day 7; n= 1, 5 | 4.0 (NA) — Standard deviation could not be calculated for CAPD cohort due to small number of participants. | -2.2 (9.78)
  Day 11; n= 1, 5: number analyzed (Participants) | 1 | 5
  Day 11; n= 1, 5 | 0.0 (NA) — Standard deviation could not be calculated for CAPD cohort due to small number of participants. | -3.2 (8.14)
  Day 17; n= 1, 4: number analyzed (Participants) | 1 | 4
  Day 17; n= 1, 4 | 5.0 (NA) — Standard deviation could not be calculated for CAPD cohort due to small number of participants. | -1.3 (13.74)

14. Secondary Outcome: Change From Baseline in Mean Corpuscular Hemoglobin Concentration (MCHC)
Description: Blood samples were collected from participants to evaluate clinical hematology parameters including MCHC. Change from Baseline in clinical hematology parameters at Day 17 are presented. Day-1 was considered as Baseline value. Change from Baseline was calculated as post-randomization values minus Baseline value. Mean and standard deviation are presented. NA indicates data is not available. Standard deviation could not be calculated for CAPD cohort due to small number of participants. Only participants with data available at the specified time point were analyzed.
Time Frame: Baseline and Day 17
Population: All Subjects Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Participants Undergoing CAPD | Participants Undergoing APD
Number analyzed (Participants) | 1 | 4
g/L | 8.0 (NA) — Standard deviation could not be calculated for CAPD cohort due to small number of participants. | 6.3 (3.86)

15. Secondary Outcome: Change From Baseline in Mean Corpuscular Volume (MCV)
Description: Blood samples were collected from participants to evaluate clinical hematology parameters including MCV. Change from Baseline in clinical hematology parameters at Day 17 are presented. Day-1 was considered as Baseline value. Change from Baseline was calculated as post-randomization values minus Baseline value. Mean and standard deviation are presented. NA indicates data is not available. Standard deviation could not be calculated for CAPD cohort due to small number of participants. Only participants with data available at the specified time point were analyzed.
Time Frame: Baseline and Day 17
Population: All Subjects Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Femtoliter
Arm/Group | Participants Undergoing CAPD | Participants Undergoing APD
Number analyzed (Participants) | 1 | 4
Femtoliter | 1.0 (NA) — Standard deviation could not be calculated for CAPD cohort due to small number of participants. | -1.5 (1.73)

16. Secondary Outcome: Change From Baseline in Mean Corpuscular Hemoglobin (MCH) Levels
Description: Blood samples were collected from participants to evaluate clinical hematology parameters including MCH. Change from Baseline in clinical hematology parameters at Day 17 are presented. Day-1 was considered as Baseline value. Change from Baseline was calculated as post-randomization values minus Baseline value. Mean and standard deviation are presented. NA indicates data is not available. Standard deviation could not be calculated for CAPD cohort due to small number of participants. Only participants with data available at the specified time point were analyzed.
Time Frame: Baseline and Day 17
Population: All Subjects Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | Participants Undergoing CAPD | Participants Undergoing APD
Number analyzed (Participants) | 1 | 4
Picograms | 1.00 (NA) — Standard deviation could not be calculated for CAPD cohort due to small number of participants. | -0.02 (0.866)

17. Secondary Outcome: Number of Participants With Abnormal Electrocardiogram (ECG) Findings
Description: Single measurements of 12-lead ECG were obtained in supine position after at least 10 minutes of rest using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT and corrected QT (QTc) interval. Participants with abnormal ECG findings at worst-case observation Carried Forward for triplicate measurements (WOCF) post-Baseline visit are presented. Only participants with data available at WOCF visit were analyzed.
Time Frame: Day 17
Population: All Subjects Population. Only those participants available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Undergoing CAPD | Participants Undergoing APD
Number analyzed (Participants) | 1 | 5
Participants | 0 | 3

18. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: Vital sign measurements including SBP and DBP were taken in a supine position after at least 5 minutes of rest. Change from Baseline in SBP and DBP at Day 17 and Day 24 (follow-up) are presented. Day-1 was considered as Baseline value. Change from Baseline was calculated as post-randomization values minus Baseline value. Mean and standard deviation are presented. NA indicates data is not available. Standard deviation could not be calculated for CAPD cohort due to small number of participants. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Baseline, Day 17 and Day 24
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Participants Undergoing CAPD | Participants Undergoing APD
Number analyzed (Participants) | 1 | 7
Millimeters of mercury
  SBP; Day 17; n= 1, 5: number analyzed (Participants) | 1 | 5
  SBP; Day 17; n= 1, 5 | 12.0 (NA) — Standard deviation could not be calculated for CAPD cohort due to small number of participants. | -10.4 (10.06)
  SBP; follow-up; n= 1, 7 | 24.0 (NA) — Standard deviation could not be calculated for CAPD cohort due to small number of participants. | -10.0 (12.46)
  DBP; Day 17; n= 1, 5: number analyzed (Participants) | 1 | 5
  DBP; Day 17; n= 1, 5 | 10.0 (NA) — Standard deviation could not be calculated for CAPD cohort due to small number of participants. | -3.4 (13.07)
  DBP; follow-up; n= 1, 7 | -4.0 (NA) — Standard deviation could not be calculated for CAPD cohort due to small number of participants. | 0.1 (12.52)

19. Secondary Outcome: Change From Baseline in Pulse Rate
Description: Vital sign measurements including pulse rate were taken in a supine position after at least 5 minutes of rest. Change from Baseline in pulse rate at Day 17 and Day 24 (follow-up) are presented. Day-1 was considered as Baseline value. Change from Baseline was calculated as post-randomization values minus Baseline value. Mean and standard deviation are presented. NA indicates data is not available. Standard deviation could not be calculated for CAPD cohort due to small number of participants. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Baseline, Day 17 and Day 24
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Participants Undergoing CAPD | Participants Undergoing APD
Number analyzed (Participants) | 1 | 7
Beats per minute
  Day 17; n= 1, 5: number analyzed (Participants) | 1 | 5
  Day 17; n= 1, 5 | -9.0 (NA) — Standard deviation could not be calculated for CAPD cohort due to small number of participants. | -5.6 (9.53)
  Follow-up; n= 1, 7 | -6.0 (NA) — Standard deviation could not be calculated for CAPD cohort due to small number of participants. | -7.0 (11.58)

20. Secondary Outcome: Change From Baseline in Body Temperature
Description: Vital sign measurements including body temperature were taken in a supine position after at least 5 minutes of rest. Change from Baseline in body temperature at Day 17 and Day 24 (follow-up) are presented. Day-1 was considered as Baseline value. Change from Baseline was calculated as post-randomization values minus Baseline value. Mean and standard deviation are presented. NA indicates data is not available. Standard deviation could not be calculated for CAPD cohort due to small number of participants. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Baseline, Day 17 and Day 24
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Degree celsius
Arm/Group | Participants Undergoing CAPD | Participants Undergoing APD
Number analyzed (Participants) | 1 | 7
Degree celsius
  Day 17; n= 1, 5: number analyzed (Participants) | 1 | 5
  Day 17; n= 1, 5 | -0.10 (NA) — Standard deviation could not be calculated for CAPD cohort due to small number of participants. | -0.20 (0.648)
  Follow-up; n= 1, 7 | -0.90 (NA) — Standard deviation could not be calculated for CAPD cohort due to small number of participants. | -0.30 (0.548)

21. Secondary Outcome: Number of Participants With Abnormal Physical Examination Findings
Description: A complete physical examination was planned to include assessments of the head, eyes, ears, nose, throat, skin, thyroid, neurological, lungs, cardiovascular, abdomen (liver and spleen), lymph nodes and extremities. This analysis was planned but not performed. Any significant finding was captured as an AE.
Time Frame: Up to Day 17
Population: All Subjects Population
Arm/Group | Participants Undergoing CAPD | Participants Undergoing APD
Number analyzed (Participants) | 0 | 0

22. Secondary Outcome: Peritoneal Dialysis Clearance of GSK1278863 and Metabolites
Description: Peritoneal dialysate samples for PK analysis of GSK1278863 and metabolites (GSK2391220, GSK2487818, GSK2506102, GSK2531398, GSK2531403 and GSK2531401) were collected. Peritoneal dialysis clearance of GSK1278863 and metabolites was calculated from Day 14 dialysate excretion data as total amount of analyte excreted over 24 hours divided by plasma AUC (0-tau). Geometric mean and geometric coefficient of variation are presented. NA indicates data is not available. Geometric coefficient of variation could not be calculated due to small number of participants. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Day 14
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Milliliter per hour
Arm/Group | Participants Undergoing CAPD | Participants Undergoing APD
Number analyzed (Participants) | 1 | 7
Milliliter per hour
  GSK1278863; n= 1, 0: number analyzed (Participants) | 1 | 0
  GSK1278863; n= 1, 0 | 12.07 (NA) — Geometric mean and geometric coefficient of variation could not be calculated for APD cohort due to insufficient data |
  GSK2391220; n= 1, 4: number analyzed (Participants) | 1 | 4
  GSK2391220; n= 1, 4 | 154.68 (NA) — Geometric mean and geometric coefficient of variation could not be calculated for APD cohort due to insufficient data | 31.68 (165.5)
  GSK2487818; n= 1, 3: number analyzed (Participants) | 1 | 3
  GSK2487818; n= 1, 3 | 124.40 (NA) — Geometric mean and geometric coefficient of variation could not be calculated for APD cohort due to insufficient data | 13.08 (195.3)
  GSK2506102; n= 1, 4: number analyzed (Participants) | 1 | 4
  GSK2506102; n= 1, 4 | 167.89 (NA) — Geometric mean and geometric coefficient of variation could not be calculated for APD cohort due to insufficient data | 40.05 (169.7)
  GSK2531398; n= 1, 4: number analyzed (Participants) | 1 | 4
  GSK2531398; n= 1, 4 | 151.29 (NA) — Geometric mean and geometric coefficient of variation could not be calculated for APD cohort due to insufficient data | 28.39 (177.5)
  GSK2531403; n= 1, 4: number analyzed (Participants) | 1 | 4
  GSK2531403; n= 1, 4 | 155.75 (NA) — Geometric mean and geometric coefficient of variation could not be calculated for APD cohort due to insufficient data | 36.18 (183.2)
  GSK2531401; n= 1, 4: number analyzed (Participants) | 1 | 4
  GSK2531401; n= 1, 4 | 201.80 (NA) — Geometric mean and geometric coefficient of variation could not be calculated for APD cohort due to insufficient data | 48.89 (199.7)

23. Secondary Outcome: Terminal Phase Half-life (t 1/2) of GSK1278863 and Metabolites
Description: Serial blood samples were collected from participants at indicated time points for PK analysis of GSK1278863 and its metabolites (GSK2391220, GSK2487818, GSK2506102, GSK2531398, GSK2531403, GSK2531401). Geometric mean and geometric coefficient of variation have been presented for all metabolites. Geometric coefficient of variation could not be calculated for CAPD cohort due to small number of participants, which is indicated by NA. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: as for outcome 1
Population: PK Population. Only participants available at specified time points were analyzed. Due to lack of quantifiable plasma concentrations in terminal elimination phase (Day 1) of 4 metabolites GSK2391220,GSK2506102,GSK2531403,GSK2531401, terminal slope(lambda z) could not be determined,thus t1/2 could not be calculated as it depends on lambda z value.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Participants Undergoing CAPD | Participants Undergoing APD
Number analyzed (Participants) | 1 | 7
Hours
  GSK1278863; Day 1; n= 1, 7 | 1.6256 (NA) — Geometric coefficient of variation could not be calculated for CAPD cohort due to small number of participants. | 1.9870 (25.8)
  GSK1278863; Day 14; n= 1, 4: number analyzed (Participants) | 1 | 4
  GSK1278863; Day 14; n= 1, 4 | 1.8088 (NA) — Geometric coefficient of variation could not be calculated for CAPD cohort due to small number of participants. | 2.5312 (35.7)
  GSK2391220; Day 14; n= 1, 4: number analyzed (Participants) | 1 | 4
  GSK2391220; Day 14; n= 1, 4 | 9.2225 (NA) — Geometric coefficient of variation could not be calculated for CAPD cohort due to small number of participants. | 10.2882 (27.2)
  GSK2487818; Day 1; n=1, 7 | 3.6560 (NA) — Geometric coefficient of variation could not be calculated for CAPD cohort due to small number of participants. | 3.3612 (22.7)
  GSK2487818; Day 14; n= 1, 4: number analyzed (Participants) | 1 | 4
  GSK2487818; Day 14; n= 1, 4 | 2.9958 (NA) — Geometric coefficient of variation could not be calculated for CAPD cohort due to small number of participants. | 3.8955 (25.3)
  GSK2506102; Day 14; n= 1,4: number analyzed (Participants) | 1 | 4
  GSK2506102; Day 14; n= 1,4 | 16.2000 (NA) — Geometric coefficient of variation could not be calculated for CAPD cohort due to small number of participants. | 17.7692 (65.4)
  GSK2531398; Day 1; n=1, 7 | 5.7900 (NA) — Geometric coefficient of variation could not be calculated for CAPD cohort due to small number of participants. | 7.0659 (35.9)
  GSK2531398; Day 14; n= 1, 4: number analyzed (Participants) | 1 | 4
  GSK2531398; Day 14; n= 1, 4 | 5.8275 (NA) — Geometric coefficient of variation could not be calculated for CAPD cohort due to small number of participants. | 7.3088 (40.0)
  GSK2531403; Day 14; n= 1, 4: number analyzed (Participants) | 1 | 4
  GSK2531403; Day 14; n= 1, 4 | 13.0606 (NA) — Geometric coefficient of variation could not be calculated for CAPD cohort due to small number of participants. | 14.5877 (43.5)
  GSK2531401; Day 14; n= 1, 4: number analyzed (Participants) | 1 | 4
  GSK2531401; Day 14; n= 1, 4 | 20.7794 (NA) — Geometric coefficient of variation could not be calculated for CAPD cohort due to small number of participants. | 26.9981 (54.2)

24. Secondary Outcome: Time of Occurrence of Cmax (Tmax) of GSK1278863 and Metabolites
Description: Serial blood samples were collected from participants at indicated time points for PK analysis of GSK1278863 and its metabolites (GSK2391220, GSK2487818, GSK2506102, GSK2531398, GSK2531403 and GSK2531401). Median and full range have been presented for all metabolites. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: Hour
Arm/Group | Participants Undergoing CAPD | Participants Undergoing APD
Number analyzed (Participants) | 1 | 7
Hour
  GSK1278863; Day 1; n=1, 7 | 0.50 [0.5 to 0.5] | 1.00 [1.0 to 3.0]
  GSK1278863; Day 14; n= 1, 4: number analyzed (Participants) | 1 | 4
  GSK1278863; Day 14; n= 1, 4 | 2.00 [2.0 to 2.0] | 2.00 [1.0 to 4.0]
  GSK2391220; Day 1; n= 1, 7 | 3.00 [3.0 to 3.0] | 4.00 [3.0 to 8.0]
  GSK2391220; Day 14; n= 1, 4: number analyzed (Participants) | 1 | 4
  GSK2391220; Day 14; n= 1, 4 | 4.00 [4.0 to 4.0] | 5.00 [4.0 to 6.0]
  GSK2487818; Day 1; n= 1, 7 | 3.00 [3.0 to 3.0] | 4.00 [2.0 to 6.0]
  GSK2487818; Day 14; n= 1, 4: number analyzed (Participants) | 1 | 4
  GSK2487818; Day 14; n= 1, 4 | 3.00 [3.0 to 3.0] | 4.00 [3.0 to 4.0]
  GSK2506102; Day 1; n=1, 7 | 4.00 [4.0 to 4.0] | 8.00 [3.0 to 12.0]
  GSK2506102; Day 14; n= 1, 4: number analyzed (Participants) | 1 | 4
  GSK2506102; Day 14; n= 1, 4 | 4.00 [4.0 to 4.0] | 5.00 [4.0 to 6.0]
  GSK2531398; Day 1; n= 1,7 | 4.00 [4.0 to 4.0] | 4.00 [3.0 to 8.0]
  GSK2531398; Day 14; n= 1, 4: number analyzed (Participants) | 1 | 4
  GSK2531398; Day 14; n= 1, 4 | 4.00 [4.0 to 4.0] | 5.00 [4.0 to 6.0]
  GSK2531403; Day 1; n= 1, 7 | 6.00 [6.0 to 6.0] | 6.00 [2.0 to 8.0]
  GSK2531403; Day 14; n= 1, 4: number analyzed (Participants) | 1 | 4
  GSK2531403; Day 14; n= 1, 4 | 4.00 [4.0 to 4.0] | 6.00 [4.0 to 6.0]
  GSK2531401; Day 1; n= 1, 7 | 8.00 [8.0 to 8.0] | 8.00 [3.0 to 12.0]
  GSK2531401; Day 14; n= 1, 4: number analyzed (Participants) | 1 | 4
  GSK2531401; Day 14; n= 1, 4 | 8.00 [8.0 to 8.0] | 9.00 [6.0 to 12.0]

25. Secondary Outcome: Accumulation Ratio of GSK1278863 and Metabolites
Description: The observed accumulation ratio was determined to estimate the extent of accumulation for GSK1278863 and metabolites (GSK2391220, GSK2487818, GSK2506102, GSK2531398, GSK2531403 and GSK2531401) after repeat dosing. Accumulation ratio was calculated by using AUC (0-tau) values at Day 1 and Day 14. Analysis was performed using mixed effect model fitted with day (single and repeat dose) as fixed effect and participant as random effect. Mean ratio and 90% confidence intervals have been presented.
Time Frame: Day 1 and Day 14
Population: PK Population. CAPD and APD arms were combined to present data for All participants analyzed.
Measure: Mean (90% Confidence Interval); unit: Ratio of AUC
Groups:
- All Participants: Participants received 1 tablet (5 mg) of GSK1278863 by oral route once daily with half glass of water for 14 days.
Arm/Group | All Participants
Number analyzed (Participants) | 8
Ratio of AUC
  GSK1278863 | 0.896 [0.645 to 1.244]
  GSK2391220 | 1.176 [1.043 to 1.326]
  GSK2487818 | 1.019 [0.944 to 1.100]
  GSK2506102 | 1.581 [1.200 to 2.081]
  GSK2531398 | 1.116 [1.015 to 1.228]
  GSK2531403 | 1.415 [1.131 to 1.771]
  GSK2531401 | 1.948 [1.301 to 2.918]

26. Secondary Outcome: Time Invariance Ratio of GSK1278863 and Metabolites
Description: Time invariance ratio for GSK1278863 and metabolites (GSK2391220, GSK2487818, GSK2506102, GSK2531398, GSK2531403 and GSK2531401) was calculated by analyzing AUC (0-inf) at Day 1 and AUC (0-tau) at Day 14. Analysis was performed using mixed effect model fitted with day (single and repeat dose) as fixed effect and participant as random effect. Mean ratio and 90% confidence intervals have been presented. NA indicates data is not available. Data could not be calculated due to insufficient data.
Time Frame: Day 1 and Day 14
Population: PK Population. CAPD and APD arms were combined to present data for all participants analyzed.
Measure: Mean (90% Confidence Interval); unit: Ratio of AUC
Arm/Group | All Participants
Number analyzed (Participants) | 8
Ratio of AUC
  GSK1278863; n= 8 | 0.896 [0.645 to 1.244]
  GSK2391220; n= 0: number analyzed (Participants) | 0
  GSK2487818; n= 8 | 1.007 [0.932 to 1.087]
  GSK2506102; n= 0: number analyzed (Participants) | 0
  GSK2531398; n= 8 | 0.986 [0.941 to 1.033]
  GSK2531403; n= 0: number analyzed (Participants) | 0
  GSK2531401; n= 0: number analyzed (Participants) | 0

27. Secondary Outcome: Plasma Concentration of Erythropoietin
Description: Serial blood samples were collected from participants at indicated time points to analyze plasma concentration of erythropoietin after repeat-dose administration of GSK1278863. Geometric mean and geometric coefficient of variation have been presented. NA indicates data is not available. Geometric coefficient of variation could not be calculated for CAPD cohort due to small number of participants. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Pre-dose and 4, 8 ,12, 24 hours post-dose on Day 1 and Day 14; Pre-dose on Day 3, 7, 11
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: IU/L
Arm/Group | Participants Undergoing CAPD | Participants Undergoing APD
Number analyzed (Participants) | 1 | 7
IU/L
  Day 1; pre-dose; n= 1, 7 | 13.860 (NA) — Geometric coefficient of variation could not be calculated for CAPD cohort due to small number of participants | 11.363 (124.9)
  Day 1; 4 hours; n= 1, 7 | 11.590 (NA) — Geometric coefficient of variation could not be calculated for CAPD cohort due to small number of participants | 14.494 (127.1)
  Day 1; 8 hours; n= 1, 7 | 23.540 (NA) — Geometric coefficient of variation could not be calculated for CAPD cohort due to small number of participants | 36.257 (96.0)
  Day 1; 12 hours; n= 1, 7 | 32.210 (NA) — Geometric coefficient of variation could not be calculated for CAPD cohort due to small number of participants | 32.629 (112.4)
  Day 1; 24 hours; n= 1, 7 | 13.570 (NA) — Geometric coefficient of variation could not be calculated for CAPD cohort due to small number of participants | 13.005 (127.5)
  Day 3; pre-dose; n= 1, 6: number analyzed (Participants) | 1 | 6
  Day 3; pre-dose; n= 1, 6 | 10.030 (NA) — Geometric coefficient of variation could not be calculated for CAPD cohort due to small number of participants | 15.452 (152.9)
  Day 7; pre-dose; n= 1, 3: number analyzed (Participants) | 1 | 3
  Day 7; pre-dose; n= 1, 3 | 5.070 (NA) — Geometric coefficient of variation could not be calculated for CAPD cohort due to small number of participants | 8.023 (66.4)
  Day 11; pre-dose; n= 1, 3: number analyzed (Participants) | 1 | 3
  Day 11; pre-dose; n= 1, 3 | 8.690 (NA) — Geometric coefficient of variation could not be calculated for CAPD cohort due to small number of participants | 9.466 (69.8)
  Day 14; pre-dose; n= 1, 4: number analyzed (Participants) | 1 | 4
  Day 14; pre-dose; n= 1, 4 | 9.490 (NA) — Geometric coefficient of variation could not be calculated for CAPD cohort due to small number of participants | 6.036 (71.2)
  Day 14; 4 hours; n= 1, 3: number analyzed (Participants) | 1 | 3
  Day 14; 4 hours; n= 1, 3 | 12.660 (NA) — Geometric coefficient of variation could not be calculated for CAPD cohort due to small number of participants | 7.674 (34.9)
  Day 14; 8 hours; n= 1, 4: number analyzed (Participants) | 1 | 4
  Day 14; 8 hours; n= 1, 4 | 30.220 (NA) — Geometric coefficient of variation could not be calculated for CAPD cohort due to small number of participants | 19.313 (81.6)
  Day 14; 12 hours; n= 1, 4: number analyzed (Participants) | 1 | 4
  Day 14; 12 hours; n= 1, 4 | 21.050 (NA) — Geometric coefficient of variation could not be calculated for CAPD cohort due to small number of participants | 25.745 (74.6)
  Day 14; 24 hours; n= 1, 4: number analyzed (Participants) | 1 | 4
  Day 14; 24 hours; n= 1, 4 | 6.590 (NA) — Geometric coefficient of variation could not be calculated for CAPD cohort due to small number of participants | 6.735 (88.1)

28. Secondary Outcome: Plasma Concentration of Hepcidin
Description: Serial blood samples were collected from participants at indicated time points to analyze plasma concentration of hepcidin after repeat-dose administration of GSK1278863. Geometric mean and geometric coefficient of variation have been presented. NA indicates data is not available. Geometric coefficient of variation could not be calculated for CAPD cohort due to small number of participants. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Pre-dose and 4, 8 ,12, 24 hours post-dose on Day 1 and Day 14; Pre-dose on Day 3, 7, 11
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per liter
Arm/Group | Participants Undergoing CAPD | Participants Undergoing APD
Number analyzed (Participants) | 1 | 7
Micrograms per liter
  Day 1; pre-dose; n= 1, 7 | 1143.00 (NA) — Geometric coefficient of variation could not be calculated for CAPD cohort due to small number of participants. | 863.21 (100.3)
  Day 1; 4 hours; n= 1, 7 | 1286.00 (NA) — Geometric coefficient of variation could not be calculated for CAPD cohort due to small number of participants. | 922.86 (108.3)
  Day 1; 8 hours; n= 1, 7 | 1427.10 (NA) — Geometric coefficient of variation could not be calculated for CAPD cohort due to small number of participants. | 760.14 (80.1)
  Day 1; 12 hours; n= 1, 7 | 1318.00 (NA) — Geometric coefficient of variation could not be calculated for CAPD cohort due to small number of participants. | 812.62 (86.1)
  Day 1; 24 hours; n= 1, 7 | 867.20 (NA) — Geometric coefficient of variation could not be calculated for CAPD cohort due to small number of participants. | 802.06 (93.5)
  Day 3; pre-dose; n= 1, 6: number analyzed (Participants) | 1 | 6
  Day 3; pre-dose; n= 1, 6 | 1021.70 (NA) — Geometric coefficient of variation could not be calculated for CAPD cohort due to small number of participants. | 819.17 (90.7)
  Day 7; pre-dose; n= 1, 4: number analyzed (Participants) | 1 | 4
  Day 7; pre-dose; n= 1, 4 | 825.30 (NA) — Geometric coefficient of variation could not be calculated for CAPD cohort due to small number of participants. | 839.42 (81.5)
  Day 11; pre-dose; n= 1, 4: number analyzed (Participants) | 1 | 4
  Day 11; pre-dose; n= 1, 4 | 852.90 (NA) — Geometric coefficient of variation could not be calculated for CAPD cohort due to small number of participants. | 800.77 (91.3)
  Day 14; pre-dose; n= 1, 4: number analyzed (Participants) | 1 | 4
  Day 14; pre-dose; n= 1, 4 | 734.30 (NA) — Geometric coefficient of variation could not be calculated for CAPD cohort due to small number of participants. | 768.33 (86.8)
  Day 14; 4 hours; n= 1, 4: number analyzed (Participants) | 1 | 4
  Day 14; 4 hours; n= 1, 4 | 847.90 (NA) — Geometric coefficient of variation could not be calculated for CAPD cohort due to small number of participants. | 782.59 (81.9)
  Day 14; 8 hours; n= 1, 4: number analyzed (Participants) | 1 | 4
  Day 14; 8 hours; n= 1, 4 | 809.90 (NA) — Geometric coefficient of variation could not be calculated for CAPD cohort due to small number of participants. | 738.96 (79.2)
  Day 14; 12 hours; n= 1, 4: number analyzed (Participants) | 1 | 4
  Day 14; 12 hours; n= 1, 4 | 705.70 (NA) — Geometric coefficient of variation could not be calculated for CAPD cohort due to small number of participants. | 757.72 (87.9)
  Day 14; 24 hours; n= 1, 4: number analyzed (Participants) | 1 | 4
  Day 14; 24 hours; n= 1, 4 | 801.30 (NA) — Geometric coefficient of variation could not be calculated for CAPD cohort due to small number of participants. | 733.66 (81.9)

ADVERSE EVENTS:
Time Frame: SAEs and non-SAEs are presented from the start of study treatment up to Day 24
Description: SAEs and non-serious AEs are reported for members of the All Subjects Population
Arm/Group | Participants Undergoing CAPD | Participants Undergoing APD
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/7
Other Adverse Events (participants affected / at risk) | 1/1 | 5/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants Undergoing CAPD (N=1) | Participants Undergoing APD (N=7)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Face oedema (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2016-06-20): https://cdn.clinicaltrials.gov/large-docs/06/NCT02243306/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-14): https://cdn.clinicaltrials.gov/large-docs/06/NCT02243306/SAP_001.pdf